CLINICAL TRIAL: NCT01530542
Title: Open-Label, Single-Dose, Randomized, 5-Period, 5-Way Crossover Study To Evaluate The Dose Proportionality And The Effects Of Food On The Bioavailability Of Acurox Tablets In Healthy Volunteers
Brief Title: A Clinical Study To Characterize The Pharmacokinetics And The Effects Of Food On Oxycodone In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: K234-10-1001; B4501006
Record Dates: First submitted 2012-01-18; First posted 2012-02-10 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Analgesia; Acute Pain; Chronic Pain; Narcotic Abuse; Opioid-related Disorders
Keywords: bioavailability; food effect; oxycodone; management of acute and chronic moderate to severe pain
MeSH Terms: conditions — Agnosia; Acute Pain; Chronic Pain; Narcotic-Related Disorders; Opioid-Related Disorders | interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment A (Experimental)
  Interventions: Drug: oxycodone hydrochloride
- Treatment B (Experimental)
  Interventions: Drug: oxycodone hydrochloride
- Treatment C (Experimental)
  Interventions: Drug: oxycodone hydrochloride
- Treatment D (Experimental)
  Interventions: Drug: oxycodone hydrochloride
- Treatment E (Experimental)
  Interventions: Drug: marketed oxycodone hydrochloride

INTERVENTIONS:
Drug: oxycodone hydrochloride — oxycodone hydrochloride 5 mg tablet under fasted conditions
  Arms: Treatment A
Drug: oxycodone hydrochloride — 2 x oxycodone hydrochloride 5 mg tablets under fasted conditions
  Arms: Treatment B
Drug: oxycodone hydrochloride — 2 x oxycodone hydrochloride 7.5 mg tablets under fasted conditions
  Arms: Treatment C
Drug: oxycodone hydrochloride — 2 x oxycodone hydrochloride 7.5 mg tablets under fed conditions
  Arms: Treatment D
Drug: marketed oxycodone hydrochloride — 1 x oxycodone hydrochloride 15 mg tablet under fed conditions
  Arms: Treatment E

SUMMARY:
This is an open-label (both the physician and healthy volunteer know which medication will be administered), single-dose, 5-dosing period study to characterize the pharmacokinetics (process by which oxycodone is absorbed, distributed, metabolized, and eliminated by the body) and the effects of food on the pharmacokinetics of oxycodone. The study will take place over approximately two and a half months and will consist of three phases: a screening visit to determine eligibility for the study, a 5-dosing period treatment phase, and an end-of-study visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between 18 and 55 years of age (inclusive)

Exclusion Criteria:

* Evidence or history of clinically significant disease;
* History of obstructive sleep apnea;
* Positive urine drug test.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2010-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, and 24 hours post-dose.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, and 24 hours post-dose.
Area under the Concentration-Time Curve (AUC) | 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, and 24 hours post-dose.
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, and 24 hours post-dose.
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] | 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, and 24 hours post-dose.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Screening up to approximately 3 months
Percentage of participants with treatment-emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) | Screening up to approximately 3 months
Change from Baseline in Diastolic Blood Pressure at each Post-Dose Assessment | 0, 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose.
Change from Baseline in Systolic Blood Pressure at each Post-Dose Assessment | 0, 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose.
Change from Baseline to each Post-Dose Assessment in Heart Rate | 0, 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose.
Change from Baseline to each Post-Dose Assessment in Respiratory Rate | 0, 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose.
Change from Baseline to each Post-Dose Assessment in Pulse Oximetry (SpO2, %) | 0, 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose.
Change from Screening to End-of-Study Assessment in Hematology Parameters | Screening up to approximately 3 months
Change from Screening to End-of-Study Assessment in Chemistry Parameters | Screening up to approximately 3 months
Change from Screening to End-of-Study Assessment in Urinalysis Parameters | Screening up to approximately 3 months
Change from Screening to End-of-Study Assessment in ECG Measurements | Screening up to approximately 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, San Antonio, Texas, United States

REFERENCES:
- [Derived] Bass A, Stark JG, Pixton GC, Sommerville KW, Zamora CA, Leibowitz M, Rolleri R. Dose proportionality and the effects of food on bioavailability of an immediate-release oxycodone hydrochloride tablet designed to discourage tampering and its relative bioavailability compared with a marketed oxycodone tablet under fed conditions: a single-dose, randomized, open-label, 5-way crossover study in healthy volunteers. Clin Ther. 2012 Jul;34(7):1601-12. doi: 10.1016/j.clinthera.2012.05.009. Epub 2012 Jun 19. PMID 22717418
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=K234-10-1001&StudyName=A%20Clinical%20Study%20To%20Characterize%20The%20Pharmacokinetics%20And%20The%20Effects%20Of%20Food%20On%20Oxycodone%20In%20Healthy%20Volunteers%0A